CLINICAL TRIAL: NCT05584787
Title: Transperineal Laser Ablation for Low and Intermediate Risk Prostate Cancer: a Single Cohort Analysis
Brief Title: Transperineal Laser Ablation for Low- and Intermediate Risk Prostate Cancer: a Single Cohort Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Carlo di Nancy Hospital (Other)
Collaborators: Elesta S.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPLA K
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; focal therapy; Echolaser; transperineal laser ablation; TPLA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPLA in patients with prostate cancer (Experimental): Patients diagnosed with low- and intermediate risk unifocal prostate cancer undergo to focal laser ablation therapy.
  Interventions: Procedure: Soractelite Echolaser Transperineal focal laser ablation

INTERVENTIONS:
Procedure: Soractelite Echolaser Transperineal focal laser ablation — US/MRI fusion laser ablation of low- and intermediate risk prostate cancer

SUMMARY:
The goal of this prospective study is to test the efficacy of Echolaser transperineal focal therapy in patients with low- and intermediate risk prostate cancer. The main question it aims to answer are: 1. short and intermediate term oncological outcomes after laser focal therapy, 2. functional outcomes and quality of life after treatment. Participants affected by low risk prostate cancer will undergo trans perineal laser focal therapy. Multiparametric prostate MRI will be perform after 3 and 12 months for oncological control. Re-fusion biopsy will be perform after 12 months. Functional outcomes and quality of life will be assess at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low- and intermediate risk prostate cancer classified as International Society for Urological Pathology, ISUP 1-2.

Exclusion Criteria:

* patients diagnosed with urothelial cancer
* contraindications for MRI
* Multifocal prostate cancer

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The trial is conducted on a population of males who underwent surgical intervention for prostate cancer.
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Oncological outcomes MRI | 3 months after treatment
  Evaluation of transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by multiparametric prostate MRI. Specifically, 1. complete ablation, 2. partial ablation or 3. persistence of cancer will be identified.
Oncological outcomes MRI | 12 months after treatment
  Evaluation of transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by multiparametric prostate MRI. Specifically, 1. complete ablation, 2. partial ablation or 3. persistence of cancer will be identified.
Oncological outcomes PSA | 3 months after treatment.
  Evaluation of transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by eventual reduction of PSA.
Oncological outcomes PSA | 6 months after treatment.
  Evaluation of transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by eventual reduction of PSA.
Oncological outcomes PSA | 12 months after treatment.
  Evaluation of transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by eventual reduction of PSA.
Oncological outcomes Re-biopsy | 12 months after treatment
  Evaluation of histological outcomes after transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by eventual negativity for cancer in a re-biopsy.

SECONDARY OUTCOMES:
Functional outcomes IPSS and IPSS QoL | 3, 6 and 12 months after treatment.
  Evaluation of lower urinary tract symptoms and quality of life after transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by the IPSS, International Prostatic Symptoms Score.
Quality of life Pain | day after surgery
  Evaluation of pain after transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by the visual analogue scale (VAS).
  The VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the parameter to be measured (pain) from 0 to 10 orientated from the left (no pain) to the right (unbearable pain).
Functional outcomes Continence | 3, 6 and 12 months after treatment.
  Evaluation of continence rate after transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by the ICIQ-SF, International Consulation on Incontinence Questionnaire - Short Form.
Functional outcomes Erection | 3, 6 and 12 months after treatment.
  Evaluation of erectile function after transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by the IIEF5, International Index of Erectile Function.
Functional outcomes Ejaculation | 3, 6 and 12 months after treatment.
  Evaluation of ejaculatory function after transperineal laser focal therapy on unifocal low- and intermediate risk prostate cancer as assessed by the MSHQ SF, Male Sexual Health Questionnaire short form.

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Bove, MD, Principal Investigator — San Carlo di Nancy Hospital
Locations (1):
- San Carlo di Nancy Hospital, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No
The analysis of the data obtained within the trial will be subject of scientific publication

REFERENCES:
- [Result] van Riel LAMJG, van Kollenburg RAA, Vis AN, van Leeuwen PJ, de Reijke TM, de Bruin DM, Oddens JR. Safety and Feasibility of Soractelite Transperineal Focal Laser Ablation for Prostate Cancer and Short-term Quality of Life Analysis from a Multicenter Pilot Study. Eur Urol Open Sci. 2022 Apr 2;39:48-54. doi: 10.1016/j.euros.2022.02.012. eCollection 2022 May. PMID 35528781